CLINICAL TRIAL: NCT00005084
Title: Pediatric Low Grade Astrocytoma: Treatment Guidance
Brief Title: Magnetic Resonance Imaging in Treating Children With Progressive Low-Grade Astrocytoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067693; UCLA-9702077; NCI-G00-1728
Record Dates: First submitted 2000-04-06; First posted 2004-06-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood low-grade cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; recurrent childhood cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Magnetic Resonance Spectroscopy; Radiotherapy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: magnetic resonance spectroscopic imaging
Radiation: radiation therapy

SUMMARY:
RATIONALE: New imaging procedures such as magnetic resonance imaging may improve the ability to determine the growth rate of progressive astrocytoma.

PURPOSE: Phase II trial to study the effectiveness of magnetic resonance imaging in treating children who have progressive low-grade astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if tumor growth rate can be decreased by targeting areas of increased choline activity, as measured by magnetic resonance spectroscopic imaging, in pediatric patients with progressive low grade astrocytoma treated with surgical resection and/or focal radiotherapy. II. Improve the quality of life without use of aggressive surgery or radiotherapy in this patient population.

OUTLINE: Patients undergo magnetic resonance spectroscopic imaging (MRSI) over 60 minutes prior to surgery and/or radiotherapy. Patients are assigned to one of two treatment arms based on tumor accessibility and may crossover to either arm. Arm I: Patients undergo conventional surgery. Arm II: Patients with inaccessible tumors undergo focal radiotherapy. Following surgery and/or radiotherapy, patients are followed every 4 months for up to 2 years with MRSI or MRI for tumor response and growth.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of low grade astrocytoma in the hypothalamus, brain stem, or thalamus of 5 cm on T2 weighted scans Incomplete surgical resection Previously treated with evidence of tumor progression No hemispheric or cerebellar masses

PATIENT CHARACTERISTICS: Age: 12 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Alger, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States